CLINICAL TRIAL: NCT01256281
Title: RESCUED: Phase I: Regional Anesthesia for Sickle Cell Crisis Using Ultrasound in The Emergency
Brief Title: Regional Anesthesia for Sickle Cell Crisis Using Ultrasound in The Emergency Department: Phase I
Acronym: RESCUED
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: lack of resources
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-0934
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Results first posted 2015-04-23 (Estimated); Last update posted 2015-04-23 (Estimated); Status verified 2015-04

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Pain; Vasoocclusion; Nerve Block; Regional Anesthesia
MeSH Terms: conditions — Anemia, Sickle Cell; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Femoral Nerve Block (Experimental): Patients enrolled will receive ultrasound guided FNB in addition to standard care. If subjects are experiencing pain in both lower extremities, both extremities will be blocked; if subjects are experiencing pain in one lower extremity, only the affected extremity will be blocked.
  Interventions: Procedure: Femoral Nerve Block

INTERVENTIONS:
Procedure: Femoral Nerve Block — Patients enrolled will receive ultrasound guided FNB in addition to standard care. If subjects are experiencing pain in both lower extremities, both extremities will be blocked; if subjects are experiencing pain in one lower extremity, only the affected extremity will be blocked.

SUMMARY:
The hypothesis of this study is:

Femoral nerve blocks can feasibly be performed on patients with Sickle Cell Disease and painful crisis in the Emergency Department.

DETAILED DESCRIPTION:
Phase I: The feasibility cohort will consist of a convenience sample. Dr. Glassberg will wear the SCD-FNB pager at all times and will enroll patients whenever logistically possible.

Participants: ED patients aged >18 who require admission for vasoocclusive pain involving the lower extremities. Vasoocclusive pain is defined as acute onset of corporeal pain, not controlled by oral analgesics, in a patient with SCD with no other apparent cause.

Description of Standard Analgesic Practices: All patients enrolled in the study will receive standardized care based on ED computer order sets designed by Drs. Shi & Glassberg and other members of the Hematology and Emergency departments (appendix E). Based on NIH52 and American Pain Society53 guidelines and current clinical evidence, these protocols were established to ensure delivery of optimal opiate therapy for patients with VOC pain. Initially, the patient will receive IV doses of opiates at the EP's discretion, followed by initiation of morphine or hydro-morphone PCA (patient controlled analgesia). PCA will continue when patient is moved to the inpatient floor, where care will also be guided by standardized order sets.

Description of the FNB Intervention: Throughout the FNB procedure, the patient will have continuous EKG, NIBP and O2 saturation monitoring. With the patient in the supine position, the leg to be blocked will be slightly abducted and externally rotated. The femoral crease and the area approximately 3 inches above and below is prepped and draped in usual sterile fashion. 1-2 ml of local anesthetic will be injected at the probable site of insertion. A sterile ultrasound probe is used to identify the femoral vessels and the femoral nerve, which usually lies 1-2 cm lateral to the artery. The femoral nerve sheath is then entered under direct visualization. Before injection, the syringe will be gently aspirated with negative blood return to ensure that the needle is not intravascular. 20mL of 0.25% bupivicaine will then be given, and deposition of anesthetic will be visualized within the nerve sheath. Intermittent aspiration and continuous ultrasound visualization during anesthetic delivery will ensure that the tip of the needle has not migrated. Injection will also be stopped and the needle repositioned if the patient complains of new or worsening pain, as this may indicate intraneural injection. If subjects are experiencing pain in both lower extremities, both extremities will be blocked; if subjects are experiencing pain in one lower extremity, only the affected extremity will be blocked.

Outcomes: This study is not exploring the efficacy of the intervention, nor is the intervention being compared to a control. Phase one is simply to verify that FNB is a feasible procedure to be performed in the ER in this population.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above
* Documented SCD: HbSS, HbSC, HbSβ0Thal, HbSβ+Thal
* Rapid onset of acute pain consistent with VOC
* Pain in at least one lower extremity
* Pain requiring admission to the hospital
* Cognitive ability to report pain on a 0-10 NRS

Exclusion Criteria:

* Primary admitting diagnosis other than VOC
* Contraindication to femoral nerve block
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey D Glassberg, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Femoral Nerve Block
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Femoral Nerve Block
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Pain Score in Legs (0-10)
Description: Pain score in legs at 2-4 hours after intervention will be the primary outcome.
  Data analysis not done.
Time Frame: 2-4 hours after intervention
Arm/Group | Femoral Nerve Block
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: there were no adverse events
Arm/Group | Femoral Nerve Block
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
study was terminated due to lack of resources. no data analysis for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes